CLINICAL TRIAL: NCT06930261
Title: Dopaminergic Disruption Induced by Traumatic Coma: Multimodal Neuroimaging Approaches to Characterize Dopaminergic Pathways Using 18F-LBT-999 PET
Brief Title: Dopaminergic Disruption Induced by Traumatic Coma: Dopaminergic Pathways Abnormalities and Biomarkers of Recovery Using MRI and 18F-LBT-999 PET
Acronym: ComaDopa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C22-62; 2023-504893-39-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-21; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-01

CONDITIONS: Coma, Traumatic
Keywords: moderate traumatic brain injury; severe traumatic brain injury
MeSH Terms: conditions — Coma, Post-Head Injury; Brain Injuries, Traumatic | interventions — 8-((E)-4-fluoro-but-2-enyl)-3beta-p-tolyl-8-aza-bicyclo(3.2.1)octane-2beta-carboxylic acid methyl ester

STUDY DESIGN:
Intervention Model Description: 3 groups:
  * Control
  * TBI-COMA (TBI with persistent coma, CGS <10, motor scale < 6)
  * TBI-REC (TBI with consciousness recovery ( i.e. response to order, GCS Motor scale =6)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TBI-COMA, TBI-REC, Control (Experimental): 18F-LBT-999 administration for all participants
  Interventions: Drug: LBT-999

INTERVENTIONS:
Drug: LBT-999 — LBT-999 administration for PET imaging

SUMMARY:
The neural correlates of consciousness have been studied at the macroscopic level. However, the neurochemical basis of these processes remains poorly understood. The mesocircuit theory challenges the cortico-centric view of consciousness. It highlights the role of subcortical regulation by dopaminergic circuits, including the ventral tegmental area and striatal loops. Experimental data show the importance of dopamine in consciousness recovery. Animal TBI studies link dopamine deficits to loss of consciousness and recovery. In humans, imaging studies show disrupted dopaminergic networks in chronic consciousness disorders. Yet, early-phase dopaminergic disruptions in acute coma remain underexplored.

Molecular imaging with PET or SPECT offers insights into dopamine system disturbances. The novel radiotracer 18F-LBT-999 enables detailed imaging of dopaminergic circuits, providing better spatial resolution and quantification than SPECT.

This proof of concept study aims to explore acute subcortical dopaminergic loop disruptions. It will combine 18F-LBT-999 PET with structural and functional MRI in post-traumatic coma.

Methods : Patients with severe traumatic brain injury (TBI) admitted to the intensive care unit state will be evaluated within 30 days post-injury. Participants will undergo clinical assessment after sedation clearance and will be categorized into three groups: (1) TBI-COMA (severe TBI with persistent coma), (2) TBI-REC (severe TBI with recovery of command-following), and (3) healthy controls. All participants will undergo clinical evaluations, anatomical and functional MRI, and molecular imaging: 18F-LBT-999-PET. Neurological outcome (CRS-r scale), Disability rating scale (DRS), Quality of life (QUOLIBRI) and axtrapyramidal symptoms (MDS-UPDRS) will be assessed at 3 month.

Primary Hypothesis: Acute post-traumatic severe TBI patients with persistent coma (TBI-COMA) show reduced presynaptic dopamine receptor levels in the striatum, compared to healthy controls.

Secondary Hypotheses:

* Dopaminergic disruptions correlate with the severity of consciousness impairment, differentiating TBI-COMA and TBI-REC groups.
* Structural damage in the striatum and nigrostriatal tract, identified via MRI, aligns with dopaminergic abnormalities.
* Multimodal imaging findings during the acute phase can predict long-term neurological and quality-of-life outcomes.
* Characterizing structural, functional, and metabolic variations in dopaminergic networks may guide personalized pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

For All Participants:

* Aged 18-65 years.
* Affiliated with or beneficiary of a social security system.
* Signed informed consent provided by the participant or a trusted representative (for patients).

For all TBI Participant

* Hospitalized for a non-penetrating traumatic brain injury (TBI) occurring within the last 30 days, with traumatic coma (Glasgow Coma Scale (GCS) < 10 and motor score (M) < 6) at hospital admission.
* Sedative treatments discontinued for more than 48 hours.
* Clinically stable (no hemodynamic, respiratory, or metabolic instability requiring specific interventions that contraindicate medical transfer to the imaging center).

For the TBI-COMA Group:

- Severe TBI characterized by prolonged coma, defined as an initial GCS < 10 with M < 6, and no recovery of consciousness at inclusion (GCS < 10 with M < 6).

For the TBI-REC Group:

* Severe TBI characterized by prolonged coma, defined as an initial GCS < 10 with M < 6, with recovery of consciousness evidenced by simple command-following (GCS ≥ 10 with M = 6) at inclusion.
* For Healthy Controls:

Matched by age (± 2 years) and sex to patients in the TBI-COMA group.

Exclusion Criteria:

For All Participants:

* Pregnant or breastfeeding women
* Contraindications to MRI
* Known allergy to the PET radiotracer or its excipients.
* History of conditions affecting the dopaminergic system
* Individuals under legal protection measures
* Current treatment with dopaminergic agonists or antagonists.

For Patients Only:

* Coma due to causes other than TBI.
* Decompressive craniectomy resulting in anatomical alterations incompatible with standardized image analysis (e.g., midline shift > 2 cm).

For Healthy Controls Only:

* Women of childbearing potential without effective contraception.
* Women unwilling to maintain effective contraception during the 30-day study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Striatal 18F-LBT-999 binding potential | 1 year after the end of inclusion
  characterization of dopaminergic network metabolic abnormalities in the TBI-COMA group. This will be assessed by comparing the binding potential (BP) of 18F-LBT-999 to presynaptic dopamine transporters in the striatum (caudate nuclei and putamen) between TBI-COMA patients and healthy controls, as measured by PET imaging

SECONDARY OUTCOMES:
Dopaminergic Network Binding (TBI-COMA vs Controls) | 1 year after the end of inclusion
  The BP of 18F-LBT-999 in dopaminergic transporters across the dopaminergic network (striatum, pallidum, substantia nigra) and brainstem (Ventral tegmental area (VTA)) will be assessed via PET in both TBI-COMA patients and healthy controls and compared between these groups
Group Comparisons (TBI-COMA vs. TBI-REC): | 1 year after the end of inclusion
  The BP of 18F-LBT-999 in the regions of interest (ROIs) described above will be compared between the TBI-COMA and TBI-REC groups
Structural and Functional Correlations | 1 year after the end of inclusion
  Relationships between dopaminergic network metabolic changes (PET) and structural or functional changes (MRI) will be explored in all TBI patients (TBI-COMA and TBI-REC):
  Metabolic Changes: BP of 18F-LBT-999 in dopaminergic network ROIs and brainstem.
  Structural White Matter Changes: Diffusion tensor imaging (DTI) tractography of nigrostriatal pathways, expressed as fractional anisotropy (FA) and mean diffusivity (MD).
  Structural Gray Matter Changes: Voxel-based morphometry (VBM) analysis in predefined ROIs and cortical regions linked to consciousness (e.g., default mode network - DMN: posterior cingulate cortex, medial prefrontal cortex), expressed as gray matter density (GMD).
  Functional Changes: Resting-state functional connectivity in the dopaminergic network and DMN, assessed via BOLD fMRI
Motor Behavioral Signatures | 1 year after the end of inclusion
  Motor behavior in TBI-COMA and TBI-REC groups will be evaluated using the Movement Disorders society- Unified Parkinson's Disease Rating Scale (MDS-UPDRS score). A 4-part scale for which the maximum score is 16 points for part 1, 52 for part 2, 108 for part 3, 23 for part 4). A higher score indicates more severe symptoms
Assessment of neurological recovery using the Coma recovery scale (CRS-R) | 3, 6 and 12 months post TBI
  Using the Coma recovery scale (CRS-R). It 's a standardized neurobehavioral assessment measure designed for use in patients with disorders of consciousness
Assessment of neurological recovery using the Disability Rating Scale (DRS) | 3, 6 and 12 months post TBI
  The Disability Rating Scale (DRS), a 30-point continuous scale that provides quantitative information to document the disability and handicap of the patient, a Higher core indicating more severe disability (i.e unresponsive wakefulness syndrome.
Measering the quality of life with the Quality of Life After Brain Injury scale (QOLIBRI). | 1 year after the end of inclusion
  This scale is made of 37 questions, assessing 6 domains of quality of life after a head injury: cognitive, affective, functional, relational, physical and emotional. The questionnaire provides a quality of life profile with a total score. A higher score indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No